CLINICAL TRIAL: NCT07251205
Title: Evaluation of a Culinary Curriculum Program for Persons Living in Recovery Residences for Opioid Use on Medication Assisted Therapy in Texas
Brief Title: Evaluating a Culinary Curriculum Program for Residents of Medication Assisted Therapy (MAT) Recovery Houses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Texas Health and Human Services Commission (Unknown)
Responsible Party: Principal Investigator, J. Michael Wilkerson, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HSC-SPH-18-0715
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Cooking Skills

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Culinary curriculum (Experimental)
  Interventions: Behavioral: Culinary curriculum

INTERVENTIONS:
Behavioral: Culinary curriculum — The curriculum has the goal of increasing nutritional knowledge and confidence in cooking skills, and it will introduce the fundamentals of cooking techniques in 5 weekly sessions. The curriculum includes introductions to cooking equipment and safety in the kitchen (basic knife skills), carbohydrate dishes, seasonal vegetables and making simple salad dressing and salads, cooking techniques (grilling, baking, and pan-frying), cooking with varying proteins, the importance of timing and organization in the kitchen, bite-size desserts, the importance of small portions, and different cultural cuisines. Additionally, the curriculum will help participants establish goals related to incorporating new ingredients.

SUMMARY:
The purpose of the study is to assess a culinary curriculum in persons with substance use disorder who are receiving medication assisted therapy and who are in recovery residences in Texas. The curriculum has the goal of increasing nutritional knowledge and confidence in cooking skills.

ELIGIBILITY:
Inclusion Criteria:

* Persons with a substance use disorder in Texas

Exclusion Criteria:

* Unable to give consent
* Does not speak English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Dietary intake as assessed by an abbreviated version of the Dietary Screener Questionnaire (DSQ) developed by the Nutrition Incentive Hub | baseline, 5 weeks
  The Abbreviated Dietary Screener Questionnaire (DSQ) asks how often in the past month different foods were eaten, for each of 9 different types of foods. For each of the 9 types of foods, data are reported categorically as follows: Never; 1 time per month; 2-3 times per month; 1 time per week ; 2 times per week; 3-4 times per week; 5-6 times per week; 1 time per day; 2 -3 times per day; 4-5 times per day; or 6 or more times per day.
Motivation to eat healthy foods as assessed by the Regulation of Eating Behavior Scale (REBS) Adapted | baseline, 5 weeks
  Total score on the Regulation of Eating Behavior Scale (REBS) Adapted ranges from 12 to 84, with a higher score indicating greater motivation to eat healthy foods.
Cooking skill self-efficacy scale as assessed by the Culinary Efficacy Scale | baseline, 5 weeks
  Total score on the Culinary Efficacy Scale ranges from 24 to 120, with a higher score indicating greater confidence in performing cooking skills.

SECONDARY OUTCOMES:
Body Mass Index (BMI) as assessed by a bioelectrical impedance analysis (BIA) device | baseline, 5 weeks
  Body mass index will be measured using a bioelectrical impedance analysis (BIA) device designed for use with children and adults.
Percent Body Fat (PBF) as assessed by a bioelectrical impedance analysis (BIA) device | baseline, 5 weeks
  Percent Body Fat (PBF) will be measured using a bioelectrical impedance analysis (BIA) device designed for use with children and adults.
Skin Carotenoid Level as assessed by the Veggie Meter | baseline, 5 weeks
  Skin Carotenoid Level will be assessed using the Veggie Meter®, which utilizes spectroscopy to quantify the concentration of carotenoids present in the skin. Carotenoids are not synthesized internally and are only obtainable through food; therefore, skin carotenoid levels can be used to detect an increase or decrease in fruit and vegetable intake over time. The VeggieMeter reports a score ranging from 0 to 800, with a higher score indicating higher skin carotenoid stores.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wilkerson, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pelletier, LG, Dion, SC, Slovinec-D'Angelo, M et al. Why Do You Regulate What You Eat? Relationships Between Forms of Regulation, Eating Behaviors, Sustained Dietary Behavior Change, and Psychological Adjustment. Motivation and Emotion. 2004; 28: 245-277.
- [Background] Condrasky MD, Williams JE, Catalano PM, Griffin SF. Development of psychosocial scales for evaluating the impact of a culinary nutrition education program on cooking and healthful eating. J Nutr Educ Behav. 2011 Nov-Dec;43(6):511-6. doi: 10.1016/j.jneb.2010.09.013. Epub 2011 Aug 15. PMID 21840764
- [Background] Karelis AD, Chamberland G, Aubertin-Leheudre M, Duval C; Ecological mobility in Aging and Parkinson (EMAP) group. Validation of a portable bioelectrical impedance analyzer for the assessment of body composition. Appl Physiol Nutr Metab. 2013 Jan;38(1):27-32. doi: 10.1139/apnm-2012-0129. Epub 2013 Jan 1. PMID 23368825
- [Background] Di Noia J, Gellermann W. Use of the Spectroscopy-Based Veggie Meter(R) to Objectively Assess Fruit and Vegetable Intake in Low-Income Adults. Nutrients. 2021 Jun 30;13(7):2270. doi: 10.3390/nu13072270. PMID 34209048
- [Background] May K, Jilcott Pitts S, Stage VC, Kelley CJ, Burkholder S, Fang X, Zeng A, Lazorick S. Use of the Veggie Meter(R) as a tool to objectively approximate fruit and vegetable intake among youth for evaluation of preschool and school-based interventions. J Hum Nutr Diet. 2020 Dec;33(6):869-875. doi: 10.1111/jhn.12755. Epub 2020 Apr 12. PMID 32281191
- See also: Nutrition Incentive Hub. (2023). Dietary Screener Questionnaire (DSQ). Dietary Screener Questionnaire (DSQ) Fruit and Vegetable Guide — https://www.nutritionincentivehub.org/resources/resource-item?resource=814e77a8-694a-455e-b28f-bb10171554a8